CLINICAL TRIAL: NCT02041897
Title: Clinical Evaluation of EUS-FNA on Diagnosis of Pancreatic Cystic Lesions----A Multiple Center,Prospective Study
Brief Title: Clinical Evaluation of EUS-FNA on Diagnosis of Pancreatic Cystic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoyin Zhang (Other)
Collaborators: Second Military Medical University (Other)
Responsible Party: Sponsor-Investigator, Xiaoyin Zhang, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCL-EUS-FNA
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cyst
Keywords: EUS-FNA; Pancreatic cystic lesion; Diagnosis
MeSH Terms: conditions — Pancreatic Cyst; Disease | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EUS-FNA, Rate of chang on diagnosis (Other): It is a single arm study. We will conclude by calculating the rate of change of diagnosis before and after getting the results of EUS-FNA.
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA — Only one puncture will be performed. First the fluid will be aspirated out for biochemical analysis and cytology. Then the tissue will be aspirated out from the solid part of the lesion for pathology.
  Other Names: Endoscopic ultrasound guided fine needle aspiration with 22G needle.

SUMMARY:
It is still controversial about the necessity of endoscopy ultrasound guide fine needle aspiration (EUS-FNA) on diagnosis of pancreatic cystic lesions(PCL).The aim of this study is to find the influence of EUS-FNA on diagnosis and suggestions of EUS specialists.

DETAILED DESCRIPTION:
First, the investigators will send only EUS images of patients with PCL to diagnosis committee that is consisted with 8 EUS specialists from different countries.The diagnosis will be collected. Then the investigators send the results of EUS-FNA. The diagnosis and suggestions will be collected again. The investigators will calculate how much diagnosis has been changed because of results of EUS-FNA. The investigators will also follow up these patients for 5 years at least to find if these patients benefit from EUS-FNA and complications such as needle tract seeding metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with ages from 18-80 years old.
2. The patients with pancreatic cystic lesions, which diameter of cystic lesion more than 2cm.
3. Sign the informed consent voluntarily. -

Exclusion Criteria:

1. The patient can't accept the endoscopic procedure.
2. The patient has blood coagulation dysfunction.
3. The patient has mental disorders.
4. The patient has mild or severe cardiorespiratory insufficiency.
5. The patient has hypertension and can't be controlled to safe level.
6. Patients with alcohol dependence.
7. Pregnant and lactating women.
8. The patients the investigators don't think suitable for this study.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Rate of change of diagnosis | During 2 weeks
  Finish diagnosis before and after getting the results of EUS-FNA

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 5 years
  after EUS-FNA

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, MD,Ph.D, Study Chair — Xijing hospital,The Fourth Military Medical University
Locations (1):
- Department of Gastroenterology,Xijing Hospital, Xian, Shanxi, China